CLINICAL TRIAL: NCT02538419
Title: Group-based Peer Support Versus Individual Education for Patients Undergoing CPAP Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Susan Redline, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014P002326
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP + Peer Support (Active Comparator): Participants randomized to this arm will receive support from a 'CPAP Peer Leader', delivered as part of a group of other participants as well as targeted one-on-one support throughout the study.
  All participants will receive CPAP in addition to this intervention.
  Interventions: Behavioral: CPAP + Peer Support
- CPAP + Individual Education (Active Comparator): Participants randomized to this arm will receive individual support and education from a trained investigator.
  All participants will receive CPAP in addition to this intervention.
  Interventions: Behavioral: CPAP + Individual Education

INTERVENTIONS:
Behavioral: CPAP + Peer Support
  Arms: CPAP + Peer Support
Behavioral: CPAP + Individual Education
  Arms: CPAP + Individual Education

SUMMARY:
The investigators will compare two alternatives designed to maximize adherence to continuous positive airway pressure (CPAP) therapy for obstructive sleep apnea (OSA) - peer-support administered in groups, versus individual education.

DETAILED DESCRIPTION:
The study is a 6-week, open-label, parallel-arm, randomized controlled trial comparing peer support and individual education (the latter of which was designed to mimic usual care). Participants in the peer-support (intervention) arm will be encouraged to attend two peer-support sessions, with one session occurring immediately prior to beginning CPAP and the other occurring two weeks later. Participants in the individual education (comparator) arm will begin CPAP without attendance at any peer-support sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with obstructive sleep apnea (no cut-off for severity)
* Prescribed continuous positive airway pressure

Exclusion Criteria:

* Not fluent in English
* Prior CPAP use at home
* Current use of any non-CPAP treatment for obstructive sleep apnea
* A co-morbid sleep disorder
* Use of supplemental oxygen
* A clinical need for urgent CPAP therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer Support: Participants randomized to this arm will receive support from a 'Peer Leader', delivered as part of a group of other participants as well as targeted one-on-one support throughout the study.
  Peer Support
- Individual Education: Participants randomized to this arm will receive individual support and education from a trained investigator.
  Individual Education
Period: Overall Study
Arm/Group | Peer Support | Individual Education
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Support | Individual Education | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (13.3) | 50.4 (13.5) | 49.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (5.3) | 30.3 (5.8) | 31.3 (6.0)
Underwent home sleep testing (as opposed to in-lab sleep testing) [Count of Participants; unit: Participants] | 16 | 16 | 32
Apnea-hypopnea index [Median (Inter-Quartile Range); unit: Events/hour] — The Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. AHI values are typically categorized as 5-15 events/hr = mild; 15-30 events/hr = moderate; and >= 30 events/h = severe
  Events/hour | 11.1 [7.6 to 25.1] | 14.3 [6.1 to 25.4] | 11.4 [7.2 to 24.6]
Oxygen saturation nadir [Median (Inter-Quartile Range); unit: % of oxygen saturation] | 81.5 [80.0 to 85.5] | 83.0 [78.0 to 87.0] | 82.5 [79.0 to 86]
Pressure 95th percentile [Median (Inter-Quartile Range); unit: cmH2O] — The 95th percentile CPAP pressure is the pressure at or below which the patient spent 95% of the time that night. Population: Two participants (intervention arm) missing data for 95th percentile pressure due to CPAP data-card error.
  cmH2O
    number analyzed (Participants) | 18 | 20 | 38
    (all) | 11.4 [10.0 to 12.1] | 10.7 [9.1 to 12.1] | 10.9 [9.2 to 12.1]
Leak 95th percentile [Median (Inter-Quartile Range); unit: liters/minute] — The 95th percentile leak is the leak level (liters/minute) at or below which the patient spent 95% of the time that night Population: Two participants (intervention arm) missing data for 95th percentile leak due to CPAP data-card error.
  liters/minute
    number analyzed (Participants) | 18 | 20 | 38
    (all) | 17.7 [5.0 to 23.7] | 17.9 [10.6 to 26.3] | 17.7 [8.1 to 24.7]
Residual apnea-hypopnea index [Median (Inter-Quartile Range); unit: events/hour] — The Apnea-hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. AHI values are typically categorized as 5-15 events/hr = mild; 15-30 events/hr = moderate; and >= 30 events/h = severe Population: Two participants (intervention arm) missing data for residual AHI due to CPAP data-card error.
  events/hour
    number analyzed (Participants) | 18 | 20 | 38
    (all) | 2.6 [0.8 to 3.6] | 2.3 [0.9 to 3.3] | 2.6 [0.8 to 3.4]
Functional Outcomes of Sleep Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Functional Outcomes of Sleep Questionnaire is a questionnaire which allows the participant to describe their sleep quality, on a scale of 5 to 20. Higher scores indicate better sleep.
  units on a scale | 16.2 (2.3) | 14.1 (3.3) | 15.2 (3.0)
Self Efficacy Measure for Sleep Apnea - Perceived Risk [Mean (Standard Deviation); unit: units on a scale] — The Self Efficacy Measure for Seep Apnea contains three sub-scales, each scored on a scale of 1 to 4. A higher score indicates a higher degree of perceived risk associated with sleep apnea.
  units on a scale | 1.5 (0.4) | 1.7 (0.4) | 1.6 (0.4)
Self Efficacy Measure for Sleep Apnea - Outcome Expectations [Mean (Standard Deviation); unit: units on a scale] — The Self Efficacy Measure for Seep Apnea contains three sub-scales, each scored on a scale of 1 to 4. A higher score indicates a higher degree of outcome expectations associated with treatment of sleep apnea.
  units on a scale | 2.0 (0.4) | 2.1 (0.6) | 2.0 (0.5)
Self Efficacy Measure for Sleep Apnea - Self Efficacy [Mean (Standard Deviation); unit: units on a scale] — The Self Efficacy Measure for Seep Apnea contains three sub-scales, each scored on a scale of 1 to 4. A higher score indicates a higher degree of self efficacy associated with treatment of sleep apnea.
  units on a scale | 2.1 (0.5) | 2.1 (0.6) | 2.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Objective adherence to CPAP, measured in hours per night.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: hours/night
Groups:
- Peer Support: Participants randomized to this arm will receive support from a 'CPAP Peer Leader', delivered as part of a group of other participants as well as targeted one-on-one support throughout the study.
  Peer Support
Arm/Group | Peer Support | Individual Education
Number analyzed (Participants) | 20 | 20
hours/night | 4.5 (2.1) | 5.0 (2.2)

2. Secondary Outcome: Percentage of Participants With Adherence >=4 Hours/Night on Average
Description: Objective adherence to CPAP, percentage with adherence >=4 hours/night on average
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peer Support | Individual Education
Number analyzed (Participants) | 20 | 20
percentage of participants | 65 | 65

3. Secondary Outcome: FOSQ
Description: Functional Outcomes of Sleep Questionnaire. The FOSQ is a questionnaire which allows the participant to describe their sleep quality, on a scale of 5 to 20. Higher scores indicate better sleep.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support | Individual Education
Number analyzed (Participants) | 20 | 20
units on a scale | 17.7 (1.3) | 16.1 (2.8)

4. Secondary Outcome: SEMSA - Perceived Risk
Description: Self Efficacy Measure for Sleep Apnea - Perceived Risk The SEMSA contains three sub-scales, each scored on a scale of 1 to 4. A higher score indicates a higher degree of perceived risk associated with sleep apnea.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support | Individual Education
Number analyzed (Participants) | 20 | 20
units on a scale | 1.6 (0.7) | 1.7 (0.6)

5. Secondary Outcome: SEMSA - Outcome Expectations
Description: Self Efficacy Measure for Sleep Apnea - Outcome Expectations. The SEMSA contains three sub-scales, each scored on a scale of 1 to 4. A higher score indicates a higher degree of outcome expectations associated with treatment of sleep apnea.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support | Individual Education
Number analyzed (Participants) | 20 | 20
units on a scale | 2.2 (0.8) | 2.3 (0.6)

6. Secondary Outcome: SEMSA - Self Efficacy
Description: Self Efficacy Measure for Sleep Apnea - Self Efficacy The SEMSA contains three sub-scales, each scored on a scale of 1 to 4. A higher score indicates a higher degree of self efficacy associated with treatment of sleep apnea.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Support | Individual Education
Number analyzed (Participants) | 20 | 20
units on a scale | 2.2 (0.8) | 2.3 (0.6)

ADVERSE EVENTS:
Arm/Group | Peer Support | Individual Education
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes